CLINICAL TRIAL: NCT00277576
Title: Phase I, Multi-Centre, Randomised, Placebo-Controlled, Dose Escalation Study to Assess Local & Systemic Tolerability of Therapeutic DNA Plasmid pdpSC18 Vaccine Administered by Particle Mediated Epidermal Delivery Using PowderJect ND10 Delivery System in Subjects With Chronic Hepatitis B Infection
Brief Title: Safety Study of HBV DNA Vaccine to Treat Patients With Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PowderMed (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PM HBV-001
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Hepatitis B
Keywords: DNA vaccine; immunotherapy; Hepatitis B Virus; Particle Mediated Epidermal Delivery
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

INTERVENTIONS:
Biological: ppdpSC18 administered by PMED

SUMMARY:
The purpose of this study is to evaluate how well the vaccine is tolerated at sites where administrations are given and any effects it may have on subjects' wellbeing. The study will also test the ability of vaccine to reduce hepatitis B disease.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is responsible for the most common form of parenterally transmitted viral hepatitis. It is estimated that approximately 350 million people worldwide are persistent carriers of the virus and it is a major cause of acute and chronic infections of the liver, with significant associated morbidity and mortality. Chronic infection occurs in 98% of new-born children infected by vertical transmission from the mother and in 5% of individuals infected after 2 years of age. About 25% of these subjects will progress to cirrhosis and 20% of this subgroup will develop hepatocellular carcinoma - one of the most common cancers world wide. HBV is a non-cytopathic virus and liver injury is mainly mediated by the host immune response against virus-infected liver cells and by the production of inflammatory cytokines. A vigorous, polyclonal and multispecific cytotoxic and helper T cell response to HBV is readily detectable in the peripheral blood of subjects with acute self-limited hepatitis B, but is weak, antigenically restricted (mono- or oligospecific) or undetectable in subjects with chronic infection. A vigorous T cell response is thus believed to be responsible for the elimination of the hepatitis B virus. The aim of a therapeutic vaccine would be to enhance natural responses by boosting the appropriate cellular immune response to HBV. The purpose of this study is to evaluate the safety and tolerability profile of the pPDPSC18 DNA vaccine as administered by Particle Mediated Epidermal Delivery (PMED )

ELIGIBILITY:
Otherwise healthy, treatment naïve subjects with chronic well compensated, eAg positive HBV infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-01; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events at all visits, vaccine site evaluations, laboratory parameters pre and post vaccination

SECONDARY OUTCOMES:
The secondary endpoints will assess the effect of the Investigational Product on:
immunological response to vaccine at each visit
clinical response to vaccine at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Henry LY Chan, Principal Investigator — Prince of Wales Hospital; Nancy Leung, Principal Investigator — Alice Ho Miu Ling Nethersole Hospital; Seng Gee Lim, Principal Investigator — National University Hospital, Singapore; Wan Cheng Chow, Principal Investigator — Singapore General Hospital; Sien-Sing Yang, Principal Investigator — Cathay General Hospital; I Shyan-Sheen, Principal Investigator — Chang Gung Memorial Hospital - Linko; Satawat Thongsawat, Principal Investigator — Maharaj Nakorn Chiang Mai Hospital; Tawesak Tandwandee, Principal Investigator — Siriraj Hospital; Man Fung Yuen, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (9):
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - 19/F Prince of Wales Hospital, Shatin
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po, N. T.
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Taiwan (2):
  - Cathay General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linko, Taoyan
- Thailand (2):
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Chiang Mai